CLINICAL TRIAL: NCT03173105
Title: Protocol Study for a Randomized Controlled Trial of the Effects of Transcranial Direct Current Stimulation (tDCS) Associated With Proprioceptive Training in Blind People
Brief Title: Effects of Transcranial Direct Current Stimulation With Proprioceptive Training in Blind People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Salgado Institute of Integral Health (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Rodolfo Borges Parreira, Rodolfo Borges Parreira, MSc, Salgado Institute of Integral Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SalgadoIIH
Record Dates: First submitted 2017-05-09; First posted 2017-06-01 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Blindness, Acquired; Blindness Congenital
Keywords: Visually Impaired Persons; Postural Balance; Rehabilitation; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Blindness | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to four groups: Group 1 (G1) - active tDCS + dynamic proprioceptive exercises; Group 2 (G2) - sham tDCS + dynamic proprioceptive exercises; Group 3 (G3)- active tDCS + static proprioceptive exercises; and Group 4 (G4) - sham tDCS + static proprioceptive exercises. Randomization will be performed with the use of sealed opaque envelopes containing a card stipulating to which group the volunteer will be allocated (G1, G2, G3 or G4).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants won´t know if they will be using the activated tDCS or Sham. The care provider also won´t know whether the participant used the tDCS or Sham as well as the outcome evaluator won´t know which is the patient´s condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (G1) (Active Comparator): active tDCS + dynamic proprioceptive exercises
  Interventions: Device: active tDCS
- Group 2 (G2) (Sham Comparator): sham tDCS + dynamic proprioceptive exercises
  Interventions: Device: sham tDCS
- Group 3 (G3) (Active Comparator): active tDCS + static proprioceptive exercises
  Interventions: Other: Dynamic proprioceptive exercises
- Group 4 (4) (Sham Comparator): sham tDCS + static proprioceptive exercises
  Interventions: Other: static proprioceptive exercises

INTERVENTIONS:
Device: active tDCS — TDCS will be administered using with two sponge (non-metallic) surface electrodes (5 x 7 cm2) moistened with saline solution. For stimulation of the motor motor, somatosensory, and visual cortices with a current of 2mA for 20 minutes. The cathode will be positioned in the medial supraorbital region.
  Other Names: tDCS - transcranial direct current stimulation
  Arms: Group 1 (G1)
Device: sham tDCS — Sham TDCS will be administered using with two sponge (non-metallic) surface electrodes (5 x 7 cm2) moistened with saline solution The stimulator will only be switched on for the first 30 seconds, giving the participant the initial sensation of tDCS, but no active stimulation throughout the remainder of the session the proprioceptive exercise session
  Other Names: tDCS - transcranial direct current stimulation
  Arms: Group 2 (G2)
Other: Dynamic proprioceptive exercises — The dynamic proprioceptive exercises will be conducted as follows: 1) walking slowly then more quickly on a trampoline; 2) walking backward with one foot behind the other; 3) walking forward on a beam; 4) going up and down a flight of stairs; and 5) sitting on a Swiss exercise ball (65 cm) and performing laterolateral, anteroposterior, circling movements and bouncing. Activities will be performed in three one-minute sets.
  Arms: Group 3 (G3)
Other: static proprioceptive exercises — The static exercises will be conducted as follows: 1) standing on toes with feet apart; and 2) with feet together; 3) standing on only right leg without support; and 4) on only left leg without support; and 5) standing with heel of right (or left) foot touching toes of left (or right) foot with feet in a straight line over on an unstable surface (wobble board) performed in six sets of 30 seconds each, with a one-minute rest interval between sets
  Arms: Group 4 (4)

SUMMARY:
Postural control requires the integration of the vestibular, visual, and somatosensory systems. Vision, in particular, exerts a considerable influence on body sway during activities that require balance. The investigators aimed to analyze the effects of transcranial direct current stimulation (tDCS) combined with proprioceptive exercises on postural control in individuals between 18 and 55 years old, with congenital and acquired blindness.

The intervention will occur in three phases: 1 - Determine differences in postural control and gait between individuals with congenital and acquired blindness with and without the use of a guide stick when wearing shoes and when barefoot; 2 - Will be a pilot study containing 10 subjects in each group (total of 40) where a sample size estimation will be analyzed based on a gait and balance parameters result from a ten consecutive days treatment protocol consisting of tDCS plus proprioceptive; 3 - A treatment protocol will be conducted in which the participants will be allocated to four groups: G1 - active tDCS + dynamic proprioceptive exercises; G2 - sham tDCS + dynamic proprioceptive exercises; G3 - active tDCS + static proprioceptive exercises; and G4 - sham tDCS + static proprioceptive exercises.

Evaluations will involve a camera system for three-dimensional gait analysis, a force plate to measure the postural control, and electromyography to analyze the muscle activities. Dynamic stability will be determined using the Timed Up and Go test and static stability will be analyzed with the aid of the force plate.

The viability of this study will allow the determination of differences in postural control between individuals with congenital and acquired blindness, the analysis of the effect of tDCS on postural control, and the establishment of a rehabilitation protocol.

DETAILED DESCRIPTION:
Ethical Aspects The study will be conducted in compliance with the principles of the Declaration of Helsinki as well as the guidelines for research involving human subjects stipulated by the National Board of Health of the Brazilian Health Ministry. Eligible individuals will receive clarifications regarding the objectives and procedures and those who agree to participate will sign a informed consentment.

Sample and recruitment The study will be conducted in three phases. First: to determine differences in postural control and gait between individuals with congenital and acquired blindness with and without a guide stick when wearing shoes and while barefoot. Second: will involve the characterization of differences in the effects of anodal tDCS on postural control and gait when stimulation is administered to different areas of the brain: primary motor cortex; somatosensory cortex; and visual cortex. Third: will involve a treatment protocol in which the participants will be randomly allocated in four groups: Group 1 - active tDCS + dynamic proprioceptive exercises; Group 2 - sham tDCS + dynamic proprioceptive exercises; Group 3 - active tDCS + static proprioceptive exercises; and Group 4 - sham tDCS + static proprioceptive exercises. Randomization will be performed with the use of sealed opaque envelopes containing a card stipulating to which group the volunteer will be allocated.

Individuals with a diagnosis of complete congenital or acquired blindness will be recruited from the community and associations that offer assistance to individuals with visual impairment. The characterization of blindness will be based on the classification of the degree of visual impairment proposed by the International Statistical Classification of Disease and the 10th Edition of the International Classification of Disease, in which visual acuity <20/400 or <20/200 in the better eye is classified as blindness.

With regard to the inclusion criteria: abnormalities of the optic nerve, retina disorders, glaucoma, Stargardt disease, macular degeneration, retinitis pigmentosa, congenital toxoplasmosis, congenital cataracts, congenital Leber's amaurosis, detached retina and astrocytoma. The exclusion criteria: medical diagnosis of injury affecting balance in the previous three years; use of medication affecting the central nervous system, coordination or balance; current symptoms of vertigo or dizziness; medical neurological diagnosis or symptoms suggestive of vestibular disorder; and past surgery or clinical condition of lower limbs or spinal column that can affect balance and gait. The subjects will be defined as independent if capable of locomotion without the assistance of others in all environments with or without the use of a guide stick.

Evaluation procedures Quantitative assessment of the gait The space-time gait parameters will be obtained with a wireless inertial detection (G-Sensor®, BTS Bioengineering SpA, Italy), previously validated in the gait assessment (Bugané et al., 2012; Pau et al., 2015).

Each sensor has 62mm × 36mm x 16mm dimensions, weighing 60g, and consists of a three-axis accelerometer (maximum scale ± 6g), a 3-axis gyroscope (full-scale ± 300°/s) and a magnetometer of 3 axes (full scale ± 6 Gauss). Data will be collected at a sampling frequency of 50Hz and will be transmitted via Bluetooth to a computer and processed using proper software of the device (BTS G-STUDIO, version: 2.6.12.0), which automatically provides the parameters (Galli et al 2015).

For data collection, participants will walk along a 15 m aisle at a self-selected speed and in a natural way. The inertia sensor will be set at the lower lumbar level (between L4-L5) with a semi-elastic belt. The device will acquire acceleration values (along three orthogonal axes: anteroposterior, mediolateral and superior-inferior) that will be transmitted via Bluetooth to a PC and processed with a software (BTS Bioengineering G-Studio®) to extract the following gait parameters: Step length; Gait speed; Cadence; Position and duration of the swing phase; Duration of the double support; Pelvic tilt.

Surface electromyography (sEMG) The sEMG analysis of the rectus femoris, tibialis anterior and soleus muscles will be performed with the aid of the eight-channel FREEEMG® electromyograph (BTS Engineering; Italy), with a bioelectric signal amplifier, wireless data transmission and bipolar electrodes with a total gain of 2000 within a frequency of 20 to 450 Hz. Impedance and the common rejection mode ratio of the equipment are >1015 Ω and 60/10 Hz 92 decibel, respectively. Electrode placement will follow the sEMG for the Non-Invasive Assessment of Muscles guidelines. All electromyographic (EMG) data will be captured and digitized in 1000 frames/second using the BTS MYOLAB® software (BTS Engineering; Italy) and will be collected simultaneously with the gait kinematics performed by the (G-Walk) and both will be managed by the BTS® system and EMG Analyzer® software, respectively.

Timed Up and Go (TUG) test This test will analyze the functional mobility and dynamic balance, in which the time (in seconds) required to stand up from a standardized chair without armrests, walk three meters, turn around, return to the chair and sit down again is recorded. The participants will be instructed to perform the test at a safe, self-selected pace. The TUG will be performed with shoes and barefoot with and without a guide stick.

Stabilometry The acquisition frequency of the force plates will be 50 Hz, captured by four piezoelectric sensors measuring 400/600 mm positioned at the extremities of each force plate. The participants will be instructed to remain in quiet standing with arms alongside the body and head held in the vertical position. Measures (45 seconds) of velocity and displacement of the center of pressure in the anteroposterior and mediolateral directions will be performed barefoot and while wearing shoes.

Intervention procedure tDCS will be administered during the therapeutic intervention sessions using the tDCS device (Trans Cranial Technologies, USA), with two sponge (non-metallic) surface electrodes measuring 5 x 7 cm2 moistened with a saline solution between 15 and 140 millimoles. The participants will be randomly allocated to two types of treatment: active and sham tDCS. Anodal tDCS will be administered over the primary motor cortex, somatosensory cortex, and the visual cortex. For stimulation of the primary motor and somatosensory cortices, the anode will be positioned over the area corresponding to the lower limbs (Cz and Pz, respectively), and the stimulation of the visual cortex, the anode will be positioned over Oz. During all three stimulations, the cathode will be positioned in the medial supraorbital region. A current of 2 milliamperes (mA) will be used for twenty minutes during each proprioceptive exercise session. For sham tDCS, the electrodes will be positioned as described, but the stimulator will only be switched on for the first 30 seconds, giving the participant the initial sensation of tDCS, but no active stimulation will be administrated throughout the remainder of the session.

Proprioceptive exercises The therapeutic intervention will be divided into static and dynamic proprioceptive exercises, which will be distributed to the groups in a random fashion. The static exercises will be conducted as follows: 1) standing on toes with feet apart; 2) standing on toes with feet together; 3) standing on only right leg without support; 4) standing on only left leg without support; and 5) standing with heel of right (or left) foot touching toes of the left (or right) foot with feet in a tandem position. The exercises will be performed on an unstable surface (wobble board) on the anteroposterior (three sets) and laterolateral (three sets) axes. Each exercise will be performed in six sets of 30 seconds each, with a one-minute rest interval between sets. The dynamic proprioceptive exercises will be conducted as follows: 1) walking slowly then more quickly on a trampoline; 2) walking backward with one foot behind the other; 3) walking forward on a beam; 4) going up and down a flight of stairs; and 5) sitting on a Swiss ball (65 cm) and performing laterolateral and anteroposterior movements, circling movements and bouncing. Activities 1 to 4 will be performed in three one-minute sets and activity five will be performed in sets with 30 seconds of each movement. Throughout all exercises, a physiotherapist will remain beside the participant to avoid excessive imbalance and the risk of falls.

Sample size estimation The sample size will be estimated from Phase II where 40 participants will be randomly allocated into four groups (10 each group). Then the calculation will be considering the minimal difference between the mean of an analysis of variance results obtained from both gait speed and the displacement of the center of pressure (COP) as the primary outcome. Thus the sample size will be estimated with a unidirectional alpha of 0.05 and an 85% statistical power. The sample determined by the calculation will be increased by 20% to compensate for possible dropouts.

Statistical analysis The data will be analyzed using the Kolmogorov-Smirnov test. Parametric variables will be expressed as mean and standard deviation. Nonparametric variables will be expressed as median and inter-quartile range. The effect size will be calculated based on the difference between means of the pre-intervention and post-intervention evaluations and will be expressed with respective 95% confidence intervals.

Analysis of variance and the Kruskal-Wallis test (nonparametric variables) will be used for the analysis of the effects obtained in the three phases of the study. The Bonferroni correction for multiple comparisons will be employed as a post hoc test. The analyses of the three phases will be performed considering spatiotemporal gait variables, Gait Variable Scores, TUG, variables related to the displacement of the center of pressure (area of displacement, displacement velocity, anteroposterior sway, and mediolateral sway) as the dependent variables. The fixed independent variables in Phase I will be group (congenital and acquired blindness) and auxiliary resource (with and without guide stick). In Phase II, the fixed independent variables will be group (tDCS over the somatosensory cortex, tDCS over the primary motor cortex and tDCS over the visual cortex) and evaluation time (pre-tDCS and post-tDCS). In Phase III, the fixed independent variables will be group (active and sham tDCS), evaluation time (pre-intervention, post-intervention and follow up), and group*evaluation time interaction. For all effects, a p-value < 0.05 will be considered indicative of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Abnormalities of the optic nerve
* Retina disorders
* Glaucoma
* Stargardt disease
* Macular degeneration
* Retinitis pigmentosa
* Congenital toxoplasmosis
* Congenital cataracts
* Congenital Leber's amaurosis
* Detached retina
* Astrocytoma

Exclusion Criteria:

* Medical diagnosis of injury affecting balance in the previous three years
* Use of medication affecting the central nervous system
* Coordination or balance
* Current symptoms of vertigo or dizziness
* Medical neurological diagnosis or symptoms suggestive of vestibular disorder
* Past surgery or clinical condition of lower limbs or spinal column that can affect balance and gait.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Postural control before and after the therapeutic proprioceptive exercises on both static and dynamic postural control in individuals with blindnes | The entire procedure will lasting about 10 minutes
  Two force plates will be used for the collection of kinematic gait data, the recording of displacement of the center of pressure and the determination of contact time between the foot and surface of the force plate

SECONDARY OUTCOMES:
Gait analysis with and without the use a guide stick, and when wearing shoes or while barefoot | For gait analysis comparison will lasting about 30 minutes
  Subjects will walk on a track five meters in lengthwhere SMART-D 140® system (BTS Engineering) will be used will be used for the collection of kinetic gait data
Surface electromyography | will lasting about 30 minutes
  The electromyographic analysis of the rectus femoris, tibialis anterior and soleum muscles will be performed with the aid of the eight-channel electromyograph. Measure will be taken during gait with and without the use a guide stick, and when wearing shoes or while barefoot
Evaluation of functional mobility | The entire procedure will lasting about 5 minutes
  Evaluation of functional mobility and dynamic balance will be performed with the Timed Up and Go Test, in which the time (seconds) required to stand up from a standardized chair without armrests, walk three meters, turn around, return to the chair and sit down again is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo B Parreira, MSc, Principal Investigator — Salgado Institute of Integral Health
Locations (1):
- Centro Universitário de Anápolis, Anápolis, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data of the variables studied such as postural control, kinematic analyzes, electromyography as well as the protocol applied to the subjects, will be available after publication of the results. Researchers may request the data from the subjects through the contact with the main investigator
Supporting Information: Study Protocol
Time Frame: all research data: informed consent, assessments, measures, and results of the given subjects will be made available immediately after publication of the study in a scientific journal
Access Criteria: Access to all information regarding the data obtained from the participants will be provided via email of the main author.

REFERENCES:
- [Background] Nashner LM, Shupert CL, Horak FB, Black FO. Organization of posture controls: an analysis of sensory and mechanical constraints. Prog Brain Res. 1989;80:411-8; discussion 395-7. doi: 10.1016/s0079-6123(08)62237-2. PMID 2699375
- [Background] Massion J. Postural control system. Curr Opin Neurobiol. 1994 Dec;4(6):877-87. doi: 10.1016/0959-4388(94)90137-6. PMID 7888772
- [Background] Rauschecker JP. Compensatory plasticity and sensory substitution in the cerebral cortex. Trends Neurosci. 1995 Jan;18(1):36-43. doi: 10.1016/0166-2236(95)93948-w. PMID 7535489
- [Background] Murnaghan CD, Squair JW, Chua R, Inglis JT, Carpenter MG. Cortical contributions to control of posture during unrestricted and restricted stance. J Neurophysiol. 2014 May;111(9):1920-6. doi: 10.1152/jn.00853.2012. Epub 2014 Feb 12. PMID 24523526
- [Background] Peterka RJ. Postural control model interpretation of stabilogram diffusion analysis. Biol Cybern. 2000 Apr;82(4):335-43. doi: 10.1007/s004220050587. PMID 10804065
- [Background] Maurer C, Peterka RJ. A new interpretation of spontaneous sway measures based on a simple model of human postural control. J Neurophysiol. 2005 Jan;93(1):189-200. doi: 10.1152/jn.00221.2004. Epub 2004 Aug 25. PMID 15331614
- [Background] Loram ID, Kelly SM, Lakie M. Human balancing of an inverted pendulum: is sway size controlled by ankle impedance? J Physiol. 2001 May 1;532(Pt 3):879-91. doi: 10.1111/j.1469-7793.2001.0879e.x. PMID 11313453
- [Background] Lesinski M, Hortobagyi T, Muehlbauer T, Gollhofer A, Granacher U. Effects of Balance Training on Balance Performance in Healthy Older Adults: A Systematic Review and Meta-analysis. Sports Med. 2015 Dec;45(12):1721-38. doi: 10.1007/s40279-015-0375-y. PMID 26325622
- [Background] Wolpert DM, Ghahramani Z, Jordan MI. An internal model for sensorimotor integration. Science. 1995 Sep 29;269(5232):1880-2. doi: 10.1126/science.7569931.
- [Background] Antal A, Kincses TZ, Nitsche MA, Paulus W. Manipulation of phosphene thresholds by transcranial direct current stimulation in man. Exp Brain Res. 2003 Jun;150(3):375-8. doi: 10.1007/s00221-003-1459-8. Epub 2003 Apr 16. PMID 12698316
- [Background] Zhou J, Hao Y, Wang Y, Jor'dan A, Pascual-Leone A, Zhang J, Fang J, Manor B. Transcranial direct current stimulation reduces the cost of performing a cognitive task on gait and postural control. Eur J Neurosci. 2014 Apr;39(8):1343-8. doi: 10.1111/ejn.12492. Epub 2014 Jan 20. PMID 24443958
- [Background] Grecco LA, de Almeida Carvalho Duarte N, Mendonca ME, Cimolin V, Galli M, Fregni F, Santos Oliveira C. Transcranial direct current stimulation during treadmill training in children with cerebral palsy: a randomized controlled double-blind clinical trial. Res Dev Disabil. 2014 Nov;35(11):2840-8. doi: 10.1016/j.ridd.2014.07.030. Epub 2014 Aug 6. PMID 25105567
- [Background] Plow EB, Obretenova SN, Fregni F, Pascual-Leone A, Merabet LB. Comparison of visual field training for hemianopia with active versus sham transcranial direct cortical stimulation. Neurorehabil Neural Repair. 2012 Jul-Aug;26(6):616-26. doi: 10.1177/1545968311431963. Epub 2012 Jan 30. PMID 22291042
- [Background] Dandona L, Dandona R. Revision of visual impairment definitions in the International Statistical Classification of Diseases. BMC Med. 2006 Mar 16;4:7. doi: 10.1186/1741-7015-4-7. PMID 16539739
- [Background] Pascolini D, Mariotti SP, Pokharel GP, Pararajasegaram R, Etya'ale D, Negrel AD, Resnikoff S. 2002 global update of available data on visual impairment: a compilation of population-based prevalence studies. Ophthalmic Epidemiol. 2004 Apr;11(2):67-115. doi: 10.1076/opep.11.2.67.28158. PMID 15255026
- [Background] Bugane F, Benedetti MG, Casadio G, Attala S, Biagi F, Manca M, Leardini A. Estimation of spatial-temporal gait parameters in level walking based on a single accelerometer: validation on normal subjects by standard gait analysis. Comput Methods Programs Biomed. 2012 Oct;108(1):129-37. doi: 10.1016/j.cmpb.2012.02.003. Epub 2012 Mar 3. PMID 22391334
- [Background] Pau M, Mandaresu S, Leban B, Nussbaum MA. Short-term effects of backpack carriage on plantar pressure and gait in schoolchildren. J Electromyogr Kinesiol. 2015 Apr;25(2):406-12. doi: 10.1016/j.jelekin.2014.11.006. Epub 2014 Dec 3. PMID 25499084
- [Result] Schmid M, Nardone A, De Nunzio AM, Schmid M, Schieppati M. Equilibrium during static and dynamic tasks in blind subjects: no evidence of cross-modal plasticity. Brain. 2007 Aug;130(Pt 8):2097-107. doi: 10.1093/brain/awm157. Epub 2007 Jul 4. PMID 17611240
- [Result] Giagazoglou P, Amiridis IG, Zafeiridis A, Thimara M, Kouvelioti V, Kellis E. Static balance control and lower limb strength in blind and sighted women. Eur J Appl Physiol. 2009 Nov;107(5):571-9. doi: 10.1007/s00421-009-1163-x. Epub 2009 Aug 22. PMID 19701648
- [Result] Choy NL, Brauer S, Nitz J. Changes in postural stability in women aged 20 to 80 years. J Gerontol A Biol Sci Med Sci. 2003 Jun;58(6):525-30. doi: 10.1093/gerona/58.6.m525. PMID 12807923
- [Result] Schwesig R, Goldich Y, Hahn A, Muller A, Kohen-Raz R, Kluttig A, Morad Y. Postural control in subjects with visual impairment. Eur J Ophthalmol. 2011 May-Jun;21(3):303-9. doi: 10.5301/EJO.2010.5504. PMID 20853264
- [Result] Sobry V, Badin P, Cernaianu S, Agnani O, Toussaint M. Do visually impaired people have a static balance as effective as sighted people? NeuroRehabilitation. 2014;35(4):851-61. doi: 10.3233/NRE-141181. PMID 25361555
- [Result] Blomqvist S, Rehn B. Validity and reliability of the dynamic one leg stance (DOLS) in people with vision loss. Advances in Physiotherapy 9(3): 129-135, 2007.
- [Result] Hakkinen A, Holopainen E, Kautiainen H, Sillanpaa E, Hakkinen K. Neuromuscular function and balance of prepubertal and pubertal blind and sighted boys. Acta Paediatr. 2006 Oct;95(10):1277-83. doi: 10.1080/08035250600573144. PMID 16982502
- [Result] Juodzbaliene V, Muckus K. The influence of the degree of visual impairment on psychomotor reaction and equilibrium maintenance of adolescents. Medicina (Kaunas). 2006;42(1):49-56. PMID 16467613
- [Result] Tomomitsu MS, Alonso AC, Morimoto E, Bobbio TG, Greve JM. Static and dynamic postural control in low-vision and normal-vision adults. Clinics (Sao Paulo). 2013 Apr;68(4):517-21. doi: 10.6061/clinics/2013(04)13. PMID 23778351
- [Result] Rubenstein LZ. Falls in older people: epidemiology, risk factors and strategies for prevention. Age Ageing. 2006 Sep;35 Suppl 2:ii37-ii41. doi: 10.1093/ageing/afl084. PMID 16926202
- [Result] Sherrington C, Tiedemann A, Fairhall N, Close JC, Lord SR. Exercise to prevent falls in older adults: an updated meta-analysis and best practice recommendations. N S W Public Health Bull. 2011 Jun;22(3-4):78-83. doi: 10.1071/NB10056. PMID 21632004
- [Result] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Result] Halko MA, Datta A, Plow EB, Scaturro J, Bikson M, Merabet LB. Neuroplastic changes following rehabilitative training correlate with regional electrical field induced with tDCS. Neuroimage. 2011 Aug 1;57(3):885-91. doi: 10.1016/j.neuroimage.2011.05.026. Epub 2011 May 18. PMID 21620985